CLINICAL TRIAL: NCT05949645
Title: Bronchoscopic Release of Air Trapped in Hyperinflated Emphysematous Lung
Brief Title: Study to Assess Safety, Feasibility, and Preliminary Efficacy of the Apreo Implant for Severe Emphysema
Acronym: BREATHE-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Apreo Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0003
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Emphysema or COPD
Keywords: hyperinflation; air-trapping; emphysema; COPD
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apreo Implant Group (Experimental): This group will undergo up to 2 procedures and will receive up to 3 implants in each lung.
  Interventions: Device: Apreo Implant Group

INTERVENTIONS:
Device: Apreo Implant Group — One or two procedures involving placement of up to three Apreo implants in the bronchial tree of each lung.

SUMMARY:
The goal of this clinical trial is to test the feasibility of an implant for severe emphysema in up to 30 participants at up to 5 study centers located in Europe and the United Kingdom. The main questions this clinical trial aim to answer are: Is it safe? Does it work?

Participants who meet eligibility criteria will have up to two procedures 30 days apart, in which up to 3 implants will be placed in each lung during the procedure(s). Participants will be asked to return for follow-up visits at 30 days, and 3, 6, and 12 months after the procedure(s).

DETAILED DESCRIPTION:
This is a first-in-human, prospective, multi-center, single-arm study assessing the safety, feasibility and preliminary efficacy of the Apreo Implant for severe emphysema in up to 30 participants. Initially all participants will undergo an Apreo Procedure involving placement of up to three implants in a native bronchial tree of one lung followed by a second Apreo Procedure 30 days later to place up to three implants in the contralateral native lung bronchial tree if indicated.

Once the fifth participant has undergone his or her first implantation procedure, implantations in currently enrolled or new participants will be paused to allow for a Safety Review Committee (SRC) to convene and review safety data once the 5th participant has completed the 7-day phone follow-up after their second Apreo Procedure (or first if only one procedure). This would be at a minimum acute procedural safety for up to 10 implantation procedures conducted in these first 5 participants, 30-day safety assessments for all 5 participants after their first lung implantations, bronchoscopic inspection 30 days after implantation of all implants in the first lung, and 7-day safety data after their first and second lung implantations. The SRC will provide comments and recommendations, including the restart of implantation for new participants, if deemed appropriate.

After the first 10 participants have completed the 7-day phone follow-up after the second Apreo Procedure (or first if only one procedure), their safety data will be reviewed by the SRC. This would include at a minimum acute procedural safety for up to 20 implantation procedures conducted in these first 10 participants, 30-day safety assessments for all 10 participants after their first lung implantations, bronchoscopic inspection 30 days after implantation of all implants in the first lung, and 7-day safety data after their first and second lung implantations. Following the review of the first 10 participants' safety data, the SRC may allow any subsequently enrolled participants to undergo one Apreo Procedure (rather than two separate procedures if appropriate for a participant) to deploy Apreo Implants in both the left and right lung airways as indicated or to continue to have all participants undergo two separate Apreo Procedures if indicated. A total of up to 30 participants will be enrolled overall.

All participants will be followed at 30 days, three, six and twelve months post the first Apreo Procedure and assessments include adverse event (AE) assessment, pulmonary function testing, bronchoscopy, and quality of life assessments (Day 30, and 3, 6, and 12 months) and an inspiratory/expiratory chest CT at 6 and 12 months. A phone follow-up for AE assessment will occur at 7 days after each Apreo Procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 35 and ≤ 80 years old
2. Computed tomography (CT) scan evidence of homogeneous or heterogeneous emphysema
3. At least one target lobe with > 35% destruction (percent of voxels with < -950 Hounsfield units on CT)
4. Post-bronchodilator ratio of FEV1/FVC < 0.7 at screening
5. Post-bronchodilator FEV1 percent predicted ≥15% and ≤50% of predicted at screening
6. Post-bronchodilator RV > 180% predicted
7. Post-bronchodilator RV/TLC ≥ 0.55 at screening
8. Marked dyspnea, scoring ≥ 2 on the modified Medical Research Council scale of 0-4
9. Cotinine testing or carboxyhemoglobin at screening indicates nonsmoker and stopped smoking at least 8 weeks before entering the trial and agrees to refrain from smoking for duration of study participation
10. Participation in a pulmonary rehabilitation program and/or confirmed to have been engaged or attempted regular physical activity in the 12 months prior to the first Apreo Procedure and agrees to continue or restart regular physical activity for the duration of the study
11. Fully vaccinated for Covid-19 (up to date per local government guidelines) and has current pneumococcus and influenza vaccination (or documented clinical intolerance)
12. Cognitively and physically able to provide written informed consent and complete participant questionnaires

Exclusion Criteria:

1. Arterial blood on room air: PaCO2 > 50 mmHg (8 kPa) or PaO2 ≤ 45 mmHg (6 kPa)
2. DLCO <20% at screening
3. Steroid therapy of 10 mg prednisolone (prednisone) or more per day
4. Two or more hospitalizations for acute exacerbations of COPD or respiratory infections in the past year before enrollment
5. Any acute exacerbation of COPD or respiratory infection less than 4 weeks before the first Apreo Procedure
6. Previous lung volume reduction surgery or lobectomy, segmentectomy or bullectomy, vapor, glue, or other pulmonary device implant
7. Known or suspected history of pulmonary arterial hypertension with a PASP > 50 mmHg on echocardiogram or mPAP > 25 mmHg on a right heart catheterization
8. Presence of a giant bulla (≥ 30% of hemithorax)
9. History of adult asthma or chronic bronchitis
10. Presence of suspicious pulmonary nodule/infiltrate that requires additional follow-up, diagnostics or treatment
11. Unequivocal and symptomatic bronchiectasis
12. Unequivocal lung cancer or other current cancer diagnosis except non-metastasized basal cell skin cancer
13. Uncontrolled hypertension (blood pressure that is inadequately treated or resistant to treatment) with a systolic > 200 mmHg or diastolic > 110 mmHg at screening or prior to first Apreo Procedure
14. Uncorrectable coagulopathy or other condition likely to increase risk of peri- or post- Apreo Procedure bleeding
15. On anticoagulant or antiplatelet therapy and unable or unwilling to hold for Apreo Procedure
16. History of myocardial infarction or unstable angina within past 6 months
17. History of a stroke less than 1 year before the first Apreo Procedure
18. Clinical history of heart failure with documented LVEF ≤ 40%
19. Clinical history of diabetes with a HbA1c > 9.0%
20. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2 (CKD-EPI) OR participant with kidney failure (Stage 5 kidney disease)
21. Mechanical ventilator dependence except participants using nocturnal bi-level positive airway pressure (biPAP) or continuous positive airway pressure (CPAP) are allowed if it would not preclude safe implantation of the study device
22. Pregnant, lactating, or women of childbearing potential who plan to become pregnant within the study duration
23. Known hypersensitivity to nitinol
24. Significantly immunocompromised, such as organ transplant recipients, those with congenital immune deficiencies, AIDS, or severe rheumatoid arthritis
25. Any disease or condition likely to limit survival to less than one year
26. Concomitant illnesses or medications that may pose a significant increased risk for complications following an Apreo Procedure
27. Currently enrolled in another trial and actively receiving experimental treatment
28. Any condition in the opinion of the investigator that would interfere with safe and complete collection of study data including the safe conduction of bronchoscopy procedures

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Serious Adverse Events (SAE) at 6 Months | 6 Months
  Rate of occurrence of serious adverse events related to the study device and/or study procedure through 6 months post-study procedure #1

SECONDARY OUTCOMES:
Device Evaluation: Device Deployment Assessment | During Procedure
  Evaluation of the ability to deploy the Apreo Implant in target airways (There is no scale - questions are assessed individually)
Device Evaluation: Device Usability Survey | During Procedure
  Evaluate operator device use challenges (There is no scale - questions are assessed individually)
Device Evaluation: Instructions for Use Survey | During Procedure
  Evaluate operator understanding of instructions for use (There is no scale - questions are assessed individually)
Efficacy Evaluation: Airway Patency at 30 Days | 30 Days
  Assess implant obstruction bronchoscopically using semi-quantitative scale (0=no narrowing of the airway to 5= >75% to 100% narrowing)
Efficacy Evaluation: Airway Patency at 3 Months | 3 Months
  Assess implant obstruction bronchoscopically using semi-quantitative scale (0=no narrowing of the airway to 5= >75% to 100% narrowing)
Efficacy Evaluation: Airway Patency at 6 Months | 6 Months
  Assess implant obstruction bronchoscopically using semi-quantitative scale (0=no narrowing of the airway to 5= >75% to 100% narrowing)
Efficacy Evaluation: Airway Patency at 12 Months | 12 Months
  Assess implant obstruction bronchoscopically using semi-quantitative scale (0=no narrowing of the airway to 5= >75% to 100% narrowing)
Efficacy Evaluation: Mucus Assessment at 30 Days | 30 Days
  Assess mucus within the Apreo Implant bronchoscopically using semi-quantitative scale (0=No mucus to 5=copious mucus)
Efficacy Evaluation: Mucus Assessment at 3 Months | 3 Months
  Assess mucus within the Apreo Implant bronchoscopically using semi-quantitative scale (0=No mucus to 5=copious mucus)
Efficacy Evaluation: Mucus Assessment at 6 Months | 6 Months
  Assess mucus within the Apreo Implant bronchoscopically using semi-quantitative scale (0=No mucus to 5=copious mucus)
Efficacy Evaluation: Mucus Assessment at 12 Months | 12 Months
  Assess mucus within the Apreo Implant bronchoscopically using semi-quantitative scale (0=No mucus to 5=copious mucus)
Efficacy Evaluation: Computed Tomography (CT) Scan at 6 Months | 6 Months
  CT evaluation of Apreo Implant diameter
Efficacy Evaluation: Computed Tomography (CT) Scan at 12 Months | 12 Months
  CT evaluation of Apreo Implant diameter
Efficacy Evaluation: Forced Expiratory Volume in 1 Second (FEV1) at 1-3 Days | 1-3 Days
  Change in FEV1 between Baseline and 1-3 days post-procedure #1
Efficacy Evaluation: Forced Expiratory Volume in 1 Second (FEV1) at 30 Days | 30 Days
  Change in FEV1 between Baseline and 30 days post-procedure #1
Efficacy Evaluation: Forced Expiratory Volume in 1 Second (FEV1) at 3 Months | 3 Months
  Change in FEV1 between Baseline and 3 months post-procedure #1
Efficacy Evaluation: Forced Expiratory Volume in 1 Second (FEV1) at 6 Months | 6 Months
  Change in FEV1 between Baseline and 6 months post-procedure #1
Efficacy Evaluation: Forced Expiratory Volume in 1 Second (FEV1) at 12 Months | 12 Months
  Change in FEV1 between Baseline and 12 months post-procedure #1
Efficacy Evaluation: Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) at 6 Months | 6 Months
  Change in DLCO between baseline and 6 months post-procedure
Efficacy Evaluation: Residual Volume (RV) at 6 Months | 6 Months
  Change in RV between baseline and 6 months as assessed by quantitative CT
Efficacy Evaluation: Residual Volume (RV) at 12 Months | 12 Months
  Change in RV between baseline and 12 months as assessed by quantitative CT
Efficacy Evaluation: Arterial Blood Gas (ABG): PaO2 at 6 Months | 6 Months
  Change in PaO2 between baseline and 6 months
Efficacy Evaluation: Arterial Blood Gas (ABG): PaCO2 at 6 Months | 6 Months
  Change in PaCO2 between baseline and 6 months
Safety: Procedural Complications | Through 24 hours post-procedure
  Percentage of participants with acute procedural complications within 24 hours of study procedure
Safety: Rate of SAEs | Through 12 Months
  Rate of occurrence of serious adverse events related to the device and/or Apreo procedure through 12 months
Safety: Rate of Adverse Device Effects | Through 12 Months
  Rate of adverse device effects through 12 months post-procedure
Efficacy Evaluation: Forced Expiratory Volume at 1 Second/ Forced Vital Capacity (FEV1/FVC) at 1-3 Days | 1-3 Days
  Change in FEV1/FVC between baseline and 1-3 days post-procedure #1
Efficacy Evaluation: Forced Expiratory Volume at 1 Second/ Forced Vital Capacity (FEV1/FVC) at 30 Days | 30 Days
  Change in FEV1/FVC between baseline and 30 days post-procedure #1
Efficacy Evaluation: Forced Expiratory Volume at 1 Second/ Forced Vital Capacity (FEV1/FVC) at 3 Months | 3 Months
  Change in FEV1/FVC between baseline and 3 months post-procedure #1
Efficacy Evaluation: Forced Expiratory Volume at 1 Second/ Forced Vital Capacity (FEV1/FVC) at 6 Months | 6 Months
  Change in FEV1/FVC between baseline and 6 months post-procedure #1
Efficacy Evaluation: Forced Expiratory Volume at 1 Second/ Forced Vital Capacity (FEV1/FVC) at 12 Months | 12 Months
  Change in FEV1/FVC between baseline and 12 months post-procedure #1
Efficacy Evaluation: Residual Volume (RV) Assessed by Pulmonary Function Testing at 1-3 Days | 1-3 Days
  Change in RV between baseline and 1-3 days
Efficacy Evaluation: Residual Volume (RV) Assessed by Pulmonary Function Testing at 30 Days | 30 Days
  Change in RV between baseline and 30 days
Efficacy Evaluation: Residual Volume (RV) Assessed by Pulmonary Function Testing at 3 Months | 3 Months
  Change in RV between baseline and 3 Months
Efficacy Evaluation: Residual Volume (RV) Assessed by Pulmonary Function Testing at 6 Months | 6 Months
  Change in RV between baseline and 6 Months
Efficacy Evaluation: Residual Volume (RV) Assessed by Pulmonary Function Testing at 12 Months | 12 Months
  Change in RV between baseline and 12 Months
Efficacy Evaluation: Residual Volume/Total Lung Capacity (RV/TLC) at 1-3 Days | 1-3 Days
  Change in RV/TLC between baseline and 1-3 days
Efficacy Evaluation: Residual Volume/Total Lung Capacity (RV/TLC) at 30 Days | 30 Days
  Change in RV/TLC between baseline and 30 days
Efficacy Evaluation: Residual Volume/Total Lung Capacity (RV/TLC) at 3 Months | 3 Months
  Change in RV/TLC between baseline and 3 months
Efficacy Evaluation: Residual Volume/Total Lung Capacity (RV/TLC) at 6 Months | 6 Months
  Change in RV/TLC between baseline and 6 months
Efficacy Evaluation: Residual Volume/Total Lung Capacity (RV/TLC) at 12 Months | 12 Months
  Change in RV/TLC between baseline and 12 months
Efficacy Evaluation: Forced Vital Capacity (FVC) at 1-3 Days | 1-3 Days
  Change in FVC between baseline and 1-3 days
Efficacy Evaluation: Forced Vital Capacity (FVC) at 30 Days | 30 Days
  Change in FVC between baseline and 30 days
Efficacy Evaluation: Forced Vital Capacity (FVC) at 3 Months | 3 Months
  Change in FVC between baseline and 3 months
Efficacy Evaluation: Forced Vital Capacity (FVC) at 6 Months | 6 Months
  Change in FVC between baseline and 6 months
Efficacy Evaluation: Forced Vital Capacity (FVC) at 12 Months | 12 Months
  Change in FVC between baseline and 12 months
Efficacy Evaluation: Six Minute Walk Test (6MWT) at 1-3 Days | 1-3 Days
  Change in 6MWT between baseline and 1-3 days
Efficacy Evaluation: Six Minute Walk Test (6MWT) at 30 Days | 30 Days
  Change in 6MWT between baseline and 30 days
Efficacy Evaluation: Six Minute Walk Test (6MWT) at 3 Months | 3 Months
  Change in 6MWT between baseline and 3 months
Efficacy Evaluation: Six Minute Walk Test (6MWT) at 6 Months | 6 Months
  Change in 6MWT between baseline and 6 months
Efficacy Evaluation: Six Minute Walk Test (6MWT) at 12 Months | 12 Months
  Change in 6MWT between baseline and 12 months
Efficacy Evaluation: Modified Borg Dyspnoea Scale at 1-3 Days | 1-3 Days
  Change in modified BORG Dyspnoea Scale between baseline and 1-3 days (scale is 0= no difficulty breathing to 10=maximal difficulty)
Efficacy Evaluation: Modified Borg Dyspnoea Scale at 30 Days | 30 Days
  Change in modified BORG Dyspnoea Scale between baseline and 30 days (scale is 0= no difficulty breathing to 10=maximal difficulty)
Efficacy Evaluation: Modified Borg Dyspnoea Scale at 3 Months | 3 Months
  Change in modified BORG Dyspnoea Scale between baseline and 3 months (scale is 0= no difficulty breathing to 10=maximal difficulty)
Efficacy Evaluation: Modified Borg Dyspnoea Scale at 6 Months | 6 Months
  Change in modified BORG Dyspnoea Scale between baseline and 6 months (scale is 0= no difficulty breathing to 10=maximal difficulty)
Efficacy Evaluation: Modified Borg Dyspnoea Scale at 12 Months | 12 Months
  Change in modified BORG Dyspnoea Scale between baseline and 12 months (scale is 0= no difficulty breathing to 10=maximal difficulty)
Efficacy Evaluation: COPD Assessment Test (CAT) at 1-3 Days (CAT scores range from 0 to 40, with higher score denoting higher impact of COPD on a participant's life) | 1-3 Days
  Change in CAT between baseline and 1-3 days
Efficacy Evaluation: COPD Assessment Test (CAT) at 30 Days (CAT scores range from 0 to 40, with higher score denoting higher impact of COPD on a participant's life) | 30 Days
  Change in CAT between baseline and 30 days
Efficacy Evaluation: COPD Assessment Test (CAT) at 3 Months (CAT scores range from 0 to 40, with higher score denoting higher impact of COPD on a participant's life) | 3 Months
  Change in CAT between baseline and 3 months
Efficacy Evaluation: COPD Assessment Test (CAT) at 6 Months (CAT scores range from 0 to 40, with higher score denoting higher impact of COPD on a participant's life) | 6 Months
  Change in CAT between baseline and 6 months
Efficacy Evaluation: COPD Assessment Test (CAT) at 12 Months (CAT scores range from 0 to 40, with higher score denoting higher impact of COPD on a participant's life) | 12 Months
  Change in CAT between baseline and 12 months
Efficacy Evaluation: St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C) at 1-3 Days (scores range from 0 to 100, with higher scores indicating more limitations to daily living) | 1-3 Days
  Change in SGRQ-C between baseline and 1-3 days
Efficacy Evaluation: St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C) at 30 Days (scores range from 0 to 100, with higher scores indicating more limitations to daily living) | 30 Days
  Change in SGRQ-C between baseline and 30 days
Efficacy Evaluation: St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C) at 3 Months (scores range from 0 to 100, with higher scores indicating more limitations to daily living) | 3 Months
  Change in SGRQ-C between baseline and 3 months
Efficacy Evaluation: St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C) at 6 Months (scores range from 0 to 100, with higher scores indicating more limitations to daily living) | 6 Months
  Change in SGRQ-C between baseline and 6 months
Efficacy Evaluation: St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C) at 12 Months (scores range from 0 to 100, with higher scores indicating more limitations to daily living) | 12 Months
  Change in SGRQ-C between baseline and 12 months
Efficacy Evaluation: Modified Medical Research Council (mMRC) Dyspnea Scale (0=no breathlessness except with strenuous exercise to 4=too breathless to leave the house or breathless when dressing or undressing) at 1-3 Days | 1-3 Days
  Change in mMRC between baseline and 1-3 days
Efficacy Evaluation: Modified Medical Research Council (mMRC) Dyspnea Scale (0=no breathlessness except with strenuous exercise to 4=too breathless to leave the house or breathless when dressing or undressing) at 30 Days | 30 Days
  Change in mMRC between baseline and 30 days
Efficacy Evaluation: Modified Medical Research Council (mMRC) Dyspnea Scale (0=no breathlessness except with strenuous exercise to 4=too breathless to leave the house or breathless when dressing or undressing) at 3 Months | 3 Months
  Change in mMRC between baseline and 3 months
Efficacy Evaluation: Modified Medical Research Council (mMRC) Dyspnea Scale (0=no breathlessness except with strenuous exercise to 4=too breathless to leave the house or breathless when dressing or undressing) at 6 Months | 6 Months
  Change in mMRC between baseline and 6 months
Efficacy Evaluation: Modified Medical Research Council (mMRC) Dyspnea Scale (0=no breathlessness except with strenuous exercise to 4=too breathless to leave the house or breathless when dressing or undressing) at 12 Months | 12 Months
  Change in mMRC between baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shirin R Hasan, Study Director — Apreo Health
Locations (3):
- Karl Landsteiner Institute, Klinik Floridsdorf, Sankt Pölten, Austria
- University Medical Center Groningen, Groningen, GZ, Netherlands
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No